CLINICAL TRIAL: NCT01224522
Title: PATIENT-MATCHED INSTRUMENTATION Versus (vs) STANDARD INSTRUMENTATION: A RANDOMIZED CLINICAL TRIAL COMPARING POSTOPERATIVE AXIAL ALIGNMENT and COMPONENT POSITION
Brief Title: Axial Alignment in Patients Operated Using the Visionaire Patient Matched Cutting Blocks
Acronym: Visionaire
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: protocol deviations
Sponsor: Smith & Nephew Orthopaedics AG (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R11025-2
Record Dates: First submitted 2010-10-14; First posted 2010-10-20 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Osteoarthritis of the Knee
Keywords: Randomized Controlled Trial; Total Knee Arthroplasty; Patient Matched Cutting Blocks
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Visionaire (Experimental): the group who will be operated by the use of Visionaire patient matched cutting blocks
  Interventions: Procedure: Visionaire
- Standard Surgical technique (Active Comparator): The group who will be operated by means fo standard surgical technique
  Interventions: Procedure: Standard surgical technique

INTERVENTIONS:
Procedure: Visionaire — Implantation of a Genesis II Total Knee by means of Visionaire patient matched cutting blocks.
  Other Names: Standard Smith & Nephew instruments; Visionaire Instruments
  Arms: Visionaire
Procedure: Standard surgical technique — Implantation of Genesis II Total Knee system by means of standard surgical technique.
  Arms: Standard Surgical technique

SUMMARY:
- Title: PATIENT-MATCHED INSTRUMENTATION VS. STANDARD INSTRUMENTATION: A RANDOMIZED CLINICAL TRIAL COMPARING POSTOPERATIVE AXIAL ALIGNMENT and COMPONENT POSITION

* Short Title: Visionaire Alignment
* Methodology: Monocentric, Single Blinded, Randomized Controlled Trial
* Study Duration: November 2010 to July 2014
* Study Centres: Leicester General Hospital, United Kingdom (UK)

DETAILED DESCRIPTION:
Malalignment is one of the main reasons for knee arthroplasty revision. With the use of patient matched cutting block we expect better axial alignment of the components.

Research Objectives:

* The primary research objective is to evaluate the axial alignment and component position in TKA with use of Smith & Nephew's VISIONAIRE Patient Matched Technology and to compare with the alignment when standard instrumentation.
* Secondary research objectives include assessing the safety and effectiveness of the VISIONAIRE patient matched technology as compared to commonly accepted standard instrumentation in patients suffering from symptomatic osteoarthritis of the knee joint.

  - Outcome Measures:
* Implant alignment and Component position by means of CT-scans
* Knee Society Score
* EuroQol-5 Dimensions (EQ-5D)
* Knee injury and Osteoarthritis Outcome Score (KOOS)
* Oxford Knee Score
* Knee-related adverse events
* Standard and full leg x-ray

  * Number of Subjects: 70 (2*35)
  * Enrollment time: 18 months
  * Diagnosis and Main Inclusion Criteria: Patients with osteoarthritis of the knee requiring total knee arthroplasty
  * Study Product, Dose, Route, Regimen:

VISIONAIRE patient matched technology versus the commonly accepted standard instrumentation for the Genesis II total knee arthroplasty implant

ELIGIBILITY:
Inclusion Criteria:

* Indication for TKA, Axial alignment between 10 degrees valgus and 20 degrees varus, BMI <36, patient must be amendable for both Genesis II total knee and Visioniare cutting blocks

Exclusion Criteria:

* Insufficient femoral or tibia bone stock, inflammatory arthritis (e.g. rheumatoid arthritis), patient is immunosuppressed, has an active infection (local or systemic), patient has physical, emotional or neurological conditions that would compromise the patients compliance with rehabilitation and follow up.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Axial Alignment | 6 weeks,
  Axial alignment will be measured by means of CT scan and long leg x-ray

SECONDARY OUTCOMES:
Clinical effectiveness and safety. | 1 year
  Safety and effectiveness will be measured by means of Knee Society Score, Oxford Score, EQ-5D and radiographic findings

CONTACTS AND LOCATIONS:
Overall Officials: Urjit Chatterji, MD, Principal Investigator — Leicester General Hospital
Locations (1):
- Leicester General Hospital, Leicester, United Kingdom